CLINICAL TRIAL: NCT07224009
Title: Phase II Clinical Trial Evaluating the Safety and Efficacy of Low Dose Naltrexone (LDN) for the Management of Fatigue in Prostate Cancer Patients on Androgen Deprivation Therapy (ADT)
Brief Title: Low Dose Naltrexone (LDN) for Management of Fatigue in Prostate Cancer Patients on Androgen Deprivation Therapy (ADT)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 299392
Record Dates: First submitted 2025-10-29; First posted 2025-11-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-arm study of low-dose naltrexone (LDN) in patients with metastatic prostate cancer, both castration-sensitive and castration-resistant, that have been on ADT for at least 3 months. Its overarching objective is to determine whether LDN can improve cancer-related fatigue and quality of life in this group of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm study of low-dose naltrexone (LDN) (Experimental): Low dose Naltrexone 3 mg is taken orally once daily to be taken with food at night. Patient will be given a pill dairy to assure compliance with the medication.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltrexone, a structurally similar compound to the opioid antagonist naloxone, but with longer half-life and higher bioavailability, was first synthesized in the 1960s and approved by Food and Drug Administration (FDA) in 1980s for treatment of opioid addiction. Its use was later expanded for management of alcohol addiction as well. The typical dose of naltrexone used for opioid and alcohol addiction is 50-100mg [19].
  Naltrexone at one-tenth of the original addiction treatment dose, referred to as LDN, exhibits interesting paradoxical pharmacology and enhances endogenous opioid production. It also showed exhibiting multiple other pharmacological effects ranging from inhibition of proliferation of cancer cells, modulating immune response there by slowing the progression of autoimmune diseases and exhibiting the inhibitory effect of pro-inflammatory cytokines thereby reducing the symptoms of neuropathic and non-cancer related pain.

SUMMARY:
The study is being done to see if a small daily dose of naltrexone (LDN, 3 mg pill) can help reduce tiredness (fatigue) in men with prostate cancer. All men in this study are being treated with hormone therapy (also called androgen deprivation therapy, or ADT). Some may also be taking newer hormone medicines such as apalutamide, daralutamide, enzalutamide, or abiraterone.

DETAILED DESCRIPTION:
The purpose of this study is to learn if low dose naltrexone can safely improve energy and reduce fatigue in men receiving these treatments.

Primary Objectives

1. Characterize mitochondrial bioenergetics, inflammation and oxidative stress after ADT and the remediating effects of LDN.
2. Assess the impact of low-dose naltrexone (LDN) on Cancer-related fatigue as measured by the FACIT-F questionnaire.

Secondary Objectives

1. Evaluate quality of life (QOL) measures [Functional Assessment of Cancer Therapy-Prostate (FACT-P) on subjects receiving LDN.
2. Evaluate safety and tolerability of LDN.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed biochemical recurrence and on ADT for at least 3 months. Metastatic castrate-sensitive and castrate-resistant prostate cancer on ADT with or without novel hormonal therapy like apalutamide, darolutamide, enzalutamide and abiraterone.
* Initiation of hormonal ablative therapy within 3 months of registration.
* ECOG performance status <3.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/μL
  * absolute neutrophil count >1,500/μL
  * platelets >100,000/μL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine ≤2.5.0
  * left ventricular ejection fraction >45%
  * FACIT-F score < 43 on screening
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Prior chemotherapy received in the last three months.
* Patients currently on PARP inhibitors.
* Currently taking or have taken within 10 days of enrollment.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Naltrexone or other agents used in the study.
* History of other malignancies other than nonmelanoma skin cancer, unless in complete remission and off therapy for that disease for at least 5 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any Patient with acute hepatitis and liver failure are excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Characterize mitochondrial bioenergetics after ADT and the remediating effects of LDN | 30 months
Characterize inflammation after ADT and the remediating effects of LDN | 30 months
Characterize oxidative stress after ADT and the remediating effects of LDN | 30 months
Assess the impact of low-dose naltrexone (LDN) on Cancer-related fatigue as measured by the FACIT-F questionnaire | 30 months

SECONDARY OUTCOMES:
Evaluate quality of life (QOL) measures [Functional Assessment of Cancer Therapy-Prostate (FACT-P) on subjects receiving LDN | 30 months
Evaluate safety and tolerability of LDN by assessing the number of participants with treatment-related adverse events graded by CTCAE v5.0 | 30 months